CLINICAL TRIAL: NCT00882791
Title: Basal Cell Carcinoma Recurrence
Brief Title: Basal Cell Carcinoma Recurrence After Mohs Surgery
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology- Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Other Study IDs: STU2538
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Basal Cell Carcinoma
Keywords: Skin Cancer; Basal Cell; Mohs surgery
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Historical Arm: 266 cases of BCC treated with Mohs surgery approximately 2-5 years ago will be assessed for recurrence.
- Prospective Arm: 300 cases of BCC will be followed annually for 3 years after Mohs surgery to assess for recurrence.

SUMMARY:
Basal cell carcinoma (BCC) is the most common skin cancer in the US and can cause significant adverse effects.

Mohs micrographic surgery, the treatment of choice for higher risk BCC, allows for removal of lesions with preservation of healthy tissue. Although the BCC recurrence rate post Mohs surgery is estimated at 1-2%, recent data is lacking to validate this historical measurement.

Our purpose is to determine the current recurrence rate of BCC after Mohs surgery.

DETAILED DESCRIPTION:
Basal cell carcinoma (BCC) is the most common nonmelanoma skin cancer in the United States, affecting nearly one million of all Americans. While BCC is rarely mortal, it has significant associated physical, psychological, and monetary costs to patients such as disfigurement and sensory loss. Individuals who have been diagnosed with at least one BCC lesion are likely to be diagnosed with more in the future. Treatment of these lesions and recurrent physician appointments can be a great inconvenience to patients, resulting in expenses to patients and loss of work and family time.

The Mohs surgery technique is associated with a low recurrence rate for BCC and is preferred for higher risk tumors and for tumors in cosmetically sensitive sites on the head and neck. While recurrence rates of BCC post Mohs are 1-2% for primary basal cells, recent data is not available to validate this historical assessment. Currently, comprehensive rates of recurrence are not available because a national registry of recurrence rates for BCC and squamous cell carcinoma (SCC) does not exist.

The purpose of this study is to both historically and prospectively assess current basal cell carcinoma recurrence rates in patients undergoing Mohs micrographic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with BCC lesions on the head, neck, genitalia, hands, or feet
* Subjects who have undergone Mohs micrographic surgery for BCC on or before December 31, 2006
* Subjects with a medical record at the respective site
* Subjects in a stable health condition, as determined by the principle investigator

Exclusion Criteria:

* Subjects with basal cell nevus syndrome
* Subjects with lesions only in areas other than the head, neck, genitalia,
* hands and feet
* Subjects who have not followed up through the Department of Dermatology
* Subjects with recurrent BCC lesions diagnosed on or prior to the recorded date of Mohs surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from Northwestern University - Department of Dermatology, Chicago, IL and from DuPage Medical Group Dermatology, Naperville, IL.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Recurrence of BCC | either after 1 study visit (historical arm), or 3 years (prospective arm)

SECONDARY OUTCOMES:
Risk Factors for recurrence of BCC | either after 1 study visit (historical arm), or 3 years (prospective arm)

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois
  - DuPage Medical Group Dermatology, Naperville, Illinois

REFERENCES:
- [Background] Mehrany K, Weenig RH, Pittelkow MR, Roenigk RK, Otley CC. High recurrence rates of Basal cell carcinoma after mohs surgery in patients with chronic lymphocytic leukemia. Arch Dermatol. 2004 Aug;140(8):985-8. doi: 10.1001/archderm.140.8.985. PMID 15313816
- [Background] Robinson JK, Fisher SG. Recurrent basal cell carcinoma after incomplete resection. Arch Dermatol. 2000 Nov;136(11):1318-24. doi: 10.1001/archderm.136.11.1318. PMID 11074691
- [Background] Dubin N, Kopf AW. Multivariate risk score for recurrence of cutaneous basal cell carcinomas. Arch Dermatol. 1983 May;119(5):373-7. PMID 6847215